CLINICAL TRIAL: NCT05475470
Title: A Prospective Randomized Controlled Trial on Safe Laparoscopic Access and Ports Insertion Using the Blade-Finger Technique
Brief Title: Blade Finger Technique for Safe Laparoscopic Entery
Acronym: new technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed lotfy, Dr, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: zuh 247
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Laparoscopic Surgery; Operative Surgical Procedure; Insufflation; Safety Issues
Keywords: veress needle; Hasson's technique; laparoscopic access; blade-finger technique

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group a (Experimental): the group we used our new blade-finger technique
  Interventions: Procedure: finger-blade technique
- group b (Experimental): the group we used Hasson's technique
  Interventions: Procedure: Hasson's technique
- group c (Experimental): the group we used veress needle technique
  Interventions: Procedure: veress needle technique

INTERVENTIONS:
Procedure: finger-blade technique — laparoscopic access technique for group a
  Other Names: laparoscopic access technique
  Arms: group a
Procedure: Hasson's technique — laparoscopic access technique for group b
  Other Names: laparoscopic access technique
  Arms: group b
Procedure: veress needle technique — laparoscopic access technique for group c
  Other Names: laparoscopic access technique for group c
  Arms: group c

SUMMARY:
blade-finger technique is a new technique for laparoscopic access which is safe

DETAILED DESCRIPTION:
after optaining irb approval and patients consented, they were divided into 3 groups to whom one of the techniques of laparoscopic entery was applied and there was a comparison between these groups

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 year-old.
* underwent laparoscopic surgery in general surgery departments in both centers from March, 2020 to May, 2022.

Exclusion Criteria:

* Patients with one or more previous abdominal surgery (upper, lower or upper and lower midline scars).
* Patients with distended abdomen due to bowel obstruction.
* Patients with uncorrected coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
time needed to access the peritoneal cavity | the first 15 minutes of operation
  the time of the procedure of access
numbers of trials till the good peritoneal access achieved | the first 15 minutes of operation
  number of trials till succeeded peritoneal access

SECONDARY OUTCOMES:
rate of complications | the first 15 minutes of operation
  bleeding, bowel injury

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided